CLINICAL TRIAL: NCT05587842
Title: Early Weightbearing vs Delayed Weightbearing After Surgical Fixation of Unstable Ankle Fractures With Syndesmosis Disruption: A Randomized Controlled Trial
Brief Title: Early vs Delayed Weightbearing After Surgical Fixation of Unstable Ankle Fractures With Syndesmosis Disruption
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Michael McKee, Professor and Chairman, Department of Orthopedic Surgery, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011244166
Record Dates: First submitted 2022-09-28; First posted 2022-10-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-12

CONDITIONS: Unstable Ankle Fractures With Syndesmotic Disruption
Keywords: Open reduction internal fixation; Syndesmotic fixation; Early weightbearing; Delayed weightbearing

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled and randomized into one of the two postoperative weightbearing groups: either the Non-weightbearing group, or the Early weightbearing.
Who Masked: Participant, Investigator
Masking Description: Allocation will be concealed to the patient and the investigators/research team until the online enrollment is completed and confirmed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-weightbearing Group (Active Comparator): At 0 weeks to 2 weeks post operation, subjects will be provided CAM (controlled ankle motion walking) boot and instructed to be non-weightbearing on the ankle, using crutches for assistance. During 2nd week, subject will visit clinic where staples/stitches will be removed, with instructions to continue non-weightbearing w/ crutches. Instructions for limited range of motion to be given, passive/active range of motion out of boot will be allowed. Between 2 to 6 weeks, the subject will continue with non-weightbearing and follow range of motion instructions. After 6 weeks, the subject will begin weightbearing as tolerated. Instructions for limited range of motion to be given, and be weaned from orthosis.
  At each follow-up visit, as part of the subject's standard of care, a physical examination and radiographic assessments will be completed, and that data collected for research purposes. Subject will also be requested to complete outcome questionnaires during their participation.
  Interventions: Procedure: Delayed Weightbearing management post operation (Traditional)
- Early weightbearing (as tolerated) Group (Experimental): At 0 weeks to 2 weeks post operation, subjects will be provided CAM (controlled ankle motion walking) boot and instructed to be non-weightbearing on the ankle, using crutches for assistance. During 2nd week, subject will visit clinic where staples/stitches will be removed, with instructions to be weightbearing as tolerated. Instructions for limited range of motion to be given, passive/active range of motion out of boot will be allowed. Between 2 to 6 weeks, subject will continue with weightbearing as tolerated in orthosis, following range of motion instructions. After 6 weeks, the subject will continue with weightbearing as tolerated, and be weaned from orthosis.
  At each follow-up visit, as part of the subject's standard of care, a physical examination and radiographic assessments will be completed, and that data collected for research purposes. Subject will also be requested to complete outcome questionnaires during their participation.
  Interventions: Procedure: Early Weightbearing management post operation

INTERVENTIONS:
Procedure: Early Weightbearing management post operation — Subjects will be instructed to be weightbearing, as tolerated, on their ankle starting at two weeks post operation.
  Arms: Early weightbearing (as tolerated) Group
Procedure: Delayed Weightbearing management post operation (Traditional) — Subjects will be instructed to be non-weightbearing on their ankle until at least 6 weeks. After 6 weeks, the subject will be instructed to be weightbearing as tolerated.
  Arms: Non-weightbearing Group

SUMMARY:
No study has prospectively compared a traditional post-operative non-weightbearing protocol versus early post-operative weightbearing as tolerated for unstable ankle injuries after surgical fixation of the syndesmosis. This prospective study will attempt to determine if early weightbearing can improve functional outcomes, result in a quicker return to work, and monitor differences in rates of adverse events. It will exclude the most severe ankle injuries and patients with excluding comorbidities.

DETAILED DESCRIPTION:
Fractures of the ankle are common injuries reported at around 10% of all fractures, with an incidence between 71-187/100,000 people/year. Rupture of the distal tibiofibular syndesmosis may occur alone or in association with ankle fractures. It is evident in approximately 10-23% of all patients with ankle fractures and approximately 20% of patients requiring internal fixation. Approximately 15/100,000 people sustain syndesmosis injuries each year, which can be associated with a variable degree of trauma to the soft-tissue and/or osseous structures that play an important role in ankle joint stability.

With syndesmotic injury, the goal of management is to restore and maintain the normal tibiofibular relationship to allow healing of the ligamentous structures of the syndesmosis. If syndesmotic injury is not detected nor treated long term, residual displacement of the ankle mortise will lead to persistent pain and early arthritis. Although most indications for surgical intervention for syndesmotic injuries are clear, certain elements of the post-operative protocol remain controversial. There is still controversy regarding using screws vs suture buttons to fix the syndesmosis, with studies showing similar functional outcomes and post-operative complications. However, screws have a significantly lower initial implant cost but inconclusive results on long term cost-effectiveness. For surgeons who use screws, two screws are better than one and recent literature shows that there is no need to remove screws routinely unless symptomatic. A recent systematic review shows there is little difference in functional outcome scores between immobilization versus early motion of surgically treated ankle fractures with syndesmotic injury. However, postoperative care in respect to when to initiate weightbearing still remains controversial.

Conventional postoperative care in regards to when to allow weightbearing varies by surgeon. Some prefer to keep the patient non-weightbearing for 6-12 weeks +/- immediate to early ankle motion, after which the patient begins protected weight bearing in a short leg walking cast for 2 weeks, followed by use of a soft ankle brace for 4-8 weeks. Others allow only touch toe weightbearing immediately postoperatively and only advance to full weight bearing once the syndesmosis screws have been removed, usually at 6 to 12 weeks. There is still no well-done evaluation to guide post op weightbearing.

A recent metanalysis of outcomes of early (EWB) versus delayed (DWB) postoperative weightbearing in patients undergoing surgical fixation of ankle fractures included seven randomized control trials, one quasi randomized trial, one prospective cohort study with retrospective matches, and one retrospective matched cohort study reported 10-point improvement in OMA scores at 6 weeks post-operatively for patients in the EWB group compared to the DWB group (p=0.02). With regards to time off work, there was a trend towards reduction of 15 days in the EWB group (p=0.08). Complication rates were similar, with no difference in rates of nonunion, malunion, or wound complications. Another systematic review does suggest that EWB after surgically treated ankle fractures would be appropriate for patients with good bone stock, minimal commination, and anatomical reduction, and may facilitate quicker rehabilitation and early return to work. Results show no significant difference in overall complication rates, including hardware failure, malunion, or nonunion. However, EWB may increase risk of superficial wound infection, but the studies had no statistical comparison.

There have been few studies to show outcomes of early protected weightbearing in patients who underwent surgical screw fixation of the syndesmosis. A recent retrospective review with 42 patients shows that EWB on a fixed syndesmosis appears to be safe, with no measurable clinical or radiographic consequences regarding ankle joint function. Even with screw breakage and loosening, loss of reduction was seldom observed. Another retrospective review was conducted on 89 patients who underwent open reduction internal fixation with syndesmotic stabilization using syndesmotic screws. The results showed maintenance of fracture reduction on all patients at 12 months and a complication rate of 11.7%, which is similar to previous early weightbearing trials on ankle fractures without syndesmotic stabilization.

No study has prospectively compared a traditional post-operative non-weightbearing protocol allowing ankle range of motion to early post-operative weightbearing as tolerated allowing ankle range of motion for unstable ankle injuries after surgical fixation of the syndesmosis. We will exclude the most severe injuries, including tibial plafond fractures with articular impaction and high-grade open ankle fractures. Implications of this study will be far reaching. Safe, early weightbearing will not only facilitate rehabilitation but it has been shown that early weightbearing reduces the time to return to work thus decreasing cost to the healthcare system and society.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ankle injury with unstable syndesmotic rupture, in the setting of isolated syndesmotic sprain, fibular fracture, bimalleolar, or trimalleolar equivalent ankle fracture
* Surgical fixation of syndesmosis and/or ankle within two weeks of injury
* Closed or low grade open (Gustilo-Anderson grade I & II low-energy injuries without gross contamination) fractures
* Skeletally mature patients with closed physis

Exclusion Criteria:

* Previous ipsilateral ankle surgery
* Bilateral ankle fractures or concurrent other lower extremity injuries/major injuries that would affect recovery time
* Inability to co-operate with post-op protocol (advanced dementia, polytrauma patient, developmental delay, etc.)
* Non-ambulatory pre-injury
* Tibial plafond fractures including articular impaction requiring elevation
* Peripheral neuropathy
* BMI over 45

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Physical Exam Functional Outcomes | Enrollment through 1 year
  Functional outcomes will be measured through physical examinations. A patients range of motion will be assessed through dorsiflexion and plantarflexion, measured from neutral ankle position, and inversion and eversion will be tested as well.
X-Ray Functional Outcomes | Enrollment through 1 year
  Additionally, functional outcomes will be assessed through x-rays. Nonunion diastasis will be defined as lack of complete cortical bridging between fragments on all radiographs. Malunion diastasis will be defined as loss of anatomic alignment on radiographs and asymmetry of the ankle clear spaces compared with the contralateral uninjured side. Symptomatic malunion diastasis will be defined as fracture union with malunion and subjective complaints including pain or instability with ambulation, weakness, fatigability, or neurologic symptoms.
Loss of reduction of the syndesmosis | Enrollment through 1 year
  Loss of reduction of the syndesmosis will be determined with radiographs that show increased tibiofibular clear space, decreased tibiofibular overlap, and/or increased medial clear space.
Olerud Molander | Enrollment through 1 year
  The Olerud score has nine categories regarding symptoms and function of the injured ankle. Patients are categorized by their individual sum scores: "poor" (0-30 points), "fair" (31-60 points.), "good" (61-90 points), and "excellent" (91-100 points).
SF36 | Enrollment through 1 year
  The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.
patient satisfaction survey | Enrollment through 1 year
  The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.

SECONDARY OUTCOMES:
Difference in rates of Adverse Events | Enrollment through 1 year
  Assessment and identification of all AEs and complications will be reported on through the data collection forms. All events will be followed from date of onset through to outcome. Type, duration, management and/or treatment of events/complications will be recorded. Those complications requiring surgical management will also be recorded on data collection forms. Patients will be closely followed during their clinical course and if a complication should arise (i.e. nonunion/malunion, infection, loss of fixation, etc.) appropriate measures, which may include re-operation, will be employed at the surgeon's discretion.

CONTACTS AND LOCATIONS:
Locations (1):
- Banner - University Medical Center, Phoenix campus, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
This information will be kept in a secure locked location. Study information will only be shared with study personnel, and the IRB and other regulatory bodies (if needed). During randomization, a subject will be assigned a unique Subject ID to maintain confidentiality.